CLINICAL TRIAL: NCT00692302
Title: Family Based Intervention for Adolescent Suicide Attempters
Brief Title: Effectiveness of a Family-Based Intervention for Adolescent Suicide Attempters (The SAFETY Study)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joan Asarnow, Professor of Psychiatry & Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH078082 (NIH); R34MH078082 (NIH); DSIR 84 CT-S
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Suicide
Keywords: Suicide Attempts; Adolescents; Suicidal; Adolescent Suicide Attempters
MeSH Terms: conditions — Suicide; Suicide, Attempted | interventions — Safety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAFETY I (Experimental): Phase I participants who will receive SAFETY
  Interventions: Behavioral: SAFETY
- SAFETY II (Experimental): Phase II participants who will receive SAFETY
  Interventions: Behavioral: SAFETY
- Control (Active Comparator): Phase II participants who will receive enhanced usual care
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: SAFETY — Participants will receive a family-based cognitive behavioral therapy intervention called SAFETY for 12 weeks. The SAFETY intervention is an individually tailored intervention strategy that integrates (1) family- and community-based interventions aimed at mobilizing family and community networks that support youth safety, adaptive behavior, and reasons for living; (2) cognitive behavioral treatment modules that focus on decreasing suicidality and preventing repeat suicide attempts; and (3) an individualized care linkage strategy that links youth to needed services and resources.
  Arms: SAFETY I; SAFETY II
Behavioral: Enhanced usual care — Enhanced usual care will include treatment as usual enhanced by study support.
  Arms: Control

SUMMARY:
This study will evaluate the effectiveness of an individually tailored suicide prevention treatment program called SAFETY in reducing suicide and suicide attempts in adolescents.

DETAILED DESCRIPTION:
Suicide is consistently a leading cause of death among adolescents in the United States, making suicide prevention a serious public health concern. The risk factors for suicide vary but are often related to depression and other mental disorders, substance abuse, a major stressful event, and family history of suicide. Despite the morbidity and mortality associated with suicide attempts in adolescents, there is a lack of empirically supported treatment strategies and consensus regarding the best practices for suicide prevention. The SAFETY intervention is an individually tailored treatment strategy that integrates family- and community-based interventions and cognitive behavioral therapy and links youth to needed services and resources. SAFETY may be an effective means of reducing suicide attempts and improving mental health in at-risk adolescents. This study will evaluate the effectiveness of SAFETY in reducing suicide and suicide attempts in adolescents.

This study will be divided into two phases. Participants in Phase I will all receive 12 weeks of the family-based cognitive behavioral therapy intervention SAFETY. Phase I will be used to develop the intervention manual, protocols, and adherence measures for SAFETY in Phase II. Phase I participants will undergo assessments at baseline and Week 12. Assessments will last 90 minutes and will include a series of interviews and questionnaires concerning family, general health, and mental health-related issues.

Participants in Phase II will be assigned randomly to receive 12 weeks of SAFETY or enhanced usual care. The frequency of sessions, which will involve both youth and parent participants, will vary on the basis of the individual needs of participants. SAFETY sessions will be individually tailored for each participant's specific needs and will include the following elements: (1) family- and community-based interventions aimed at mobilizing family and community networks that support youth safety, adaptive behavior, and reasons for living; (2) cognitive behavioral treatment modules that focus on decreasing suicidality and preventing repeat suicide attempts; and (3) an individualized care linkage strategy that links youth to needed services and resources. At baseline, Week 12, and Month 6, all youth and parent participants will undergo the same assessments that were performed during Phase I.

ELIGIBILITY:
Inclusion Criteria:

* Suicide attempt or repetitive self-harm in the 3 months before study entry

Exclusion Criteria:

* Psychosis
* Substance dependency
* Immediate risk of out-of-home placement
* Symptoms/conditions that would interfere with assessment and/or intervention protocols

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Suicide Attempt | 3-months
  Derived from adapted C-SSRS that incorporates questions from the Suicide History Interview
Suicide-related hospitalizations | Measured at month 3
  SACA, adapted

OTHER OUTCOMES:
Suicide Attempts | 3-months
  Derived from adapted C-SSRS that incorporates questions from the Suicide History Interview
Suicide-related hospitalizations | 3-months
  SACA, adapted
Suicide-related ED Visits | 3-Months
  SACA, adapted
Suicide-related ED visits | Final assessment
  SACA, adapted
Youth Depression | 3-months
  CES-D
Youth Hopelessness | 3-months
  BHS
Parent Depression | 3 Months
  CES-D
Parent Hopelessness | 3 Months
  BHS
Youth Suicidality (Ideation and Behavior) | 3 months
  HASS
Youth Social Adjustment | 3 months
  SAS-SR for Youth

CONTACTS AND LOCATIONS:
Overall Officials: Joan R. Asarnow, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, California, United States

REFERENCES:
- [Result] Asarnow JR, Hughes JL, Babeva KN, Sugar CA. Cognitive-Behavioral Family Treatment for Suicide Attempt Prevention: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2017 Jun;56(6):506-514. doi: 10.1016/j.jaac.2017.03.015. Epub 2017 Apr 5. PMID 28545756
- [Result] Asarnow JR, Berk M, Hughes JL, Anderson NL. The SAFETY Program: a treatment-development trial of a cognitive-behavioral family treatment for adolescent suicide attempters. J Clin Child Adolesc Psychol. 2015;44(1):194-203. doi: 10.1080/15374416.2014.940624. Epub 2014 Sep 25. PMID 25255931
- [Result] Babeva KN, Klomhaus AM, Sugar CA, Fitzpatrick O, Asarnow JR. Adolescent Suicide Attempt Prevention: Predictors of Response to a Cognitive-Behavioral Family and Youth Centered Intervention. Suicide Life Threat Behav. 2020 Feb;50(1):56-71. doi: 10.1111/sltb.12573. Epub 2019 Jul 26. PMID 31350782
- See also: Center for Trauma-Informed Adolescent Suicide, Self-harm & Substance Abuse Treatment & Prevention — http://www.asapnctsn.org